CLINICAL TRIAL: NCT02906436
Title: Pilot Study of Lung Transplantation After Ex-Vivo Lung Reconditioning
Brief Title: Ex-Vivo Lung Reconditioning
Acronym: ExVivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/36; 2010-A00879-30 (Other: ANSM)
Record Dates: First submitted 2016-09-11; First posted 2016-09-20 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Lung Transplantation
Keywords: Lung transplantation; ExVivo reconditionning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ExVivo lung reconditioning (Experimental)
  Interventions: Device: Xvivo Chamber

INTERVENTIONS:
Device: Xvivo Chamber

SUMMARY:
Only about 15% of the potential candidates for lung donation are considered suitable for transplantation. Thus, a strategy that could improve the quality and precision of assessment of nonacceptable donor lungs could have a major impact on reducing waiting time and mortality while on the list.

A new method for ex vivo lung perfusion (EVLP) has been developed recently by Steen and colleagues to assess the quality of lungs from a non-heart-beating donor. The method can also be used to recondition "marginal" and nonacceptable donor lungs.

After harvesting, the lungs were perfused ex vivo with Steen Solution, an extracellular matrix with high colloid osmotic pressure. A membrane oxygenator connected to the circuit received gas from a mixture of nitrogen and carbon dioxide, maintaining a normal mixed venous blood gas level in the perfusate. The lungs were gradually rewarmed, reperfused, and ventilated for evaluation through analyses of oxygenation capacity, pulmonary vascular resistance (PVR), lung compliance (LC), and biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the waiting list for lung transplantation and for which the Biomedicine -Agency has awarded a lung transplantation after Ex-Vivo lung reconditioning
* Patients affiliated to a social security system;
* Patients who consented to participate in writing

Exclusion Criteria:

-Patients under tutorship or unable to consent or institutionalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
number of "transplantable" grafts and Reduced waiting time before transplantation | 12 months

SECONDARY OUTCOMES:
Difference of data obtained 2 hours after Ex-Vivo lung reconditioning with those obtained 4 hours after Ex-Vivo lung reconditioning | 4 hours after Ex-Vivo lung reconditioning
Number of deaths of patients on waiting list | 5 years
survival time after lung transplantation with ExVivo lung reconditioning | 1 year after end of study
Quality of life scale score after lung transplantation with ExVivo lung reconditioning | 1 year after end of study

CONTACTS AND LOCATIONS:
Overall Officials: Alain Chapelier, PhD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - Centre chirugical Marie Lannelongue, Le Plessis-Robinson
  - Hopital Foch, Suresnes